CLINICAL TRIAL: NCT03225274
Title: "A Study to Evaluate the Effectiveness of Breathing Exercises as Therapeutic Play on Respiratory Status Among Children Undergoing Nebulization Therapy With Lower Respiratory Tract Disorders in Selected Hospitals of Haryana."
Brief Title: Effectiveness of Breathing Exercises as Therapeutic Play on Respiratory Status Among Children With Lower Respiratory Tract Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, shally chaudhary, student, MSc. Nursing, Maharishi Markendeswar University (Deemed to be University)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 778
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Respiratory Status
Keywords: Breathing exercises; Respiratory status; Nebulization therapy; lower respiratory tract disorders
MeSH Terms: interventions — Breathing Exercises; Play Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Experimental Group consist of 30 subjects. Pre-assessment of respiratory status among children was assessed. Then after 5 minutes of administration of Nebulization, breathing exercises as therapeutic play (balloon inflation, candle blowing, blow air into water with a straw was administered for 15 minutes once in a day for 3 days consecutively and then post-assessment was taken daily 5 minutes after the administration of breathing exercises as therapeutic play.
  Interventions: Other: Breathing Exercises as Therapeutic Play
- Comparison Group (No Intervention): Comparison Group consist of 30 subjects. Pre-assessment of respiratory status among children was assessed. Then only nebulization therapy was administered and then post-assessment was taken daily after 25 minutes of administered.

INTERVENTIONS:
Other: Breathing Exercises as Therapeutic Play — On day 1, pre- intervention assessment of respiratory status was done before administration of breathing exercises as therapeutic play and after 5 minutes of administration of Nebulization therapy, breathing exercises was administered among children for 15 minutes once in a day and then after 5 minutes 1st post-intervention assessment was done on same day.
  On 2nd day again after 5 minutes of administration of Nebulization therapy, breathing exercises was administered among children for 15 minutes once in a day and after 5 minutes again post-intervention assessment was done on same day.
  On 3rd day again after 5 minutes of administration of Nebulization therapy, breathing exercises was administered among children for 15 minutes once in a day and after 5 minutes again post-intervention assessment was done on same day.
  Arms: Experimental Group

SUMMARY:
The study evaluates the effectiveness of Breathing Exercises as Therapeutic Play on respiratory Status among children with Lower respiratory Tract Disorders. patient were allocated into two groups- Experimental group and Comparison group. Experimental Group received Breathing Exercises as Therapeutic Play after administration of Nebulization therapy and comparison Group received no Breathing Exercises.

DETAILED DESCRIPTION:
The subjects were selected by Purposive sampling technique and allocated into 2 groups i.e experimental and comparison group. the total sample size for the study was 60 children i.e 30 in Experiment Group and 30 in Comparison group.

Experimental Group- Pre-assessment of respiratory status among children was assessed. Then after 5 minutes of administration of Nebulization, breathing exercises as therapeutic play (balloon inflation, candle blowing, blow air into water with a straw was administered for 15 minutes once in a day for 3 days consecutively and then post-assessment was taken daily 5 minutes after the administration of breathing exercises as therapeutic play.

Comparison Group- Pre-assessment of respiratory status among children was assessed. Then only nebulization therapy was administered and then post-assessment was taken daily after 25 minutes of administered.

ELIGIBILITY:
Inclusion Criteria:

* 5-18 years of age
* prescribed with Nebulization therapy
* able to understand hindi.
* available during the period of data collection and willing to participate in study.

Exclusion Criteria:

* having upper respiratory tract infection
* on ventilator support.
* coming to hospital for OPD visits.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Modified Clinical Respiratory Score | 10 minutes
  To assess the Respiratory Status of children. The scoring of Modified Clinical Respiratory Score from 0 (Mild Respiratory status) to 12(Severe respiratory status)

CONTACTS AND LOCATIONS:
Overall Officials: Mr. Yogesh Kumar, M.Sc Nursing, Study Director — Maharishi Markandeshwar University

REFERENCES:
- [Background] Nair H, Nokes DJ, Gessner BD, Dherani M, Madhi SA, Singleton RJ, O'Brien KL, Roca A, Wright PF, Bruce N, Chandran A, Theodoratou E, Sutanto A, Sedyaningsih ER, Ngama M, Munywoki PK, Kartasasmita C, Simoes EA, Rudan I, Weber MW, Campbell H. Global burden of acute lower respiratory infections due to respiratory syncytial virus in young children: a systematic review and meta-analysis. Lancet. 2010 May 1;375(9725):1545-55. doi: 10.1016/S0140-6736(10)60206-1. PMID 20399493
- [Background] Acharya D, Prasanna KS, Nair S, Rao RS. Acute respiratory infections in children: a community based longitudinal study in south India. Indian J Public Health. 2003 Jan-Mar;47(1):7-13. PMID 14723289